CLINICAL TRIAL: NCT01733056
Title: Characterization of Immune Response to Vaccination in Patients Receiving Single-Drug Immunosuppressive Therapy
Brief Title: Immune Response to Vaccination in Patients Receiving Single Drug Immunosuppression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Robert A Swerlick MD, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00044264; 5-31040 (Other Grant/Funding Number: Emory U19 grant Award account number 5-31040)
Record Dates: First submitted 2012-11-20; First posted 2012-11-26 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-06

CONDITIONS: Immunosuppression
Keywords: Dermatology; Influenza Vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy Volunteer (Placebo Comparator): Healthy volunteers without skin disease that received administration of Fluzone
  Interventions: Biological: Flu Vaccine
- Azathioprine (Experimental): Patients with skin diseases taking azathioprine that received administration of Fluzone
  Interventions: Biological: Flu Vaccine
- TNF alpha blocker (Experimental): Patients with skin diseases taking azathioprine that received administration of Fluzone
  Interventions: Biological: Flu Vaccine

INTERVENTIONS:
Biological: Flu Vaccine — Administration of Fluzone (Influenza Vaccine)

SUMMARY:
Biomedical Lay Summary Title: Characterization of immune response to vaccination in patients receiving single-drug immunosuppressive therapy Principal Investigator: Robert Swerlick, MD Other Investigators: Rafi Ahmed, PhD Suephy Chen, MD Jens Wrammert, PhD Adam Sperduto

1. Problem of Interest We are proposing to study the effectiveness of vaccines in people who are taking drugs that affect the immune system. There are many populations of people who have chronic medical conditions that require them to have long-term treatment with immunosuppressive medications (drugs that decrease the function of the immune system). Examples of these patients include organ transplant recipients, patients with immune cell cancers such as leukemia and lymphoma, patients with inflammatory disorders such as lupus or scleroderma, and patients with skin conditions requiring steroid-based creams, ointments, pills, or injections. Patients who are taking these medications should receive appropriate vaccinations such as tetanus boosters, influenza vaccines, and pneumonia vaccines. The effectiveness of vaccinations depends in large part on a strong response to the vaccine by the immune system. Drugs that decrease immune system function therefore, may also decrease the effectiveness of vaccines.
2. How the Problem of Interest will be studied

We plan to give three different groups of participants influenza vaccinations and measure each participant's immune system response through blood tests. The three groups will be:

1. Healthy people taking no immunosuppressive medications
2. Patients with skin conditions requiring treatment with azathioprine and currently taking no other immunosuppressive agents
3. Patients with psoriasis requiring treatment with TNF-alpha (tumor necrosis factor-alpha) and currently taking no other immunosuppressive medications.

All participants will be between 18 - 89 years old and will not have had influenza vaccination within the previous six months. We will administer the vaccination on day 0. We will take blood samples on days 0, 7, and 28 following vaccination. We will use these blood samples to measure the amount of antibodies produced to the vaccine and the response of specific immune system cells known as B-lymphocytes. Using statistical methods, we will compare these findings between the three groups of participants to determine if differences in response to the vaccination exist.

3. How the research will advance scientific knowledge and/or human health To our knowledge there is no scientific data available regarding the effectiveness of vaccinations in patients receiving only one specific immunosuppressive medication. We will also be using new techniques developed at Emory to measure the B-lymphocyte response to the vaccine. This research could potentially help guide vaccination strategies for people requiring immunosuppressive medications and prevent infectious disease in these populations as well as the general population.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 89 years of age
* Patient Taking azathioprine, Humira, Enbrel or Remicade
* Willing to participate in the healthy volunteer arm

Exclusion Criteria:

* Has received flu vaccine in past year
* Taking systemic corticosteroids or any other immunosuppressive drug

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Swerlick, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University, Department of Dermatology, Atlanta, Georgia
  - Emory University, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 43 subjects enrolled from Dept of dermatology, including 21 normal controls, 12 patients on TNF blockers for the treatment of skin diseases, and 10 patients treated with azathioprine for the treatment of skin diseases. Both serologic and cell based assays were completed before and after vaccination on all subjects.
Period: Overall Study
Arm/Group | Healthy Volunteer | Azathioprine | TNF Alpha Blockers
Started | 21 | 10 | 12
Completed | 21 | 10 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Volunteer: Healthy volunteers without skin disease prior to influenza vaccination
- Azathioprine: Patients with skin diseases taking azathioprine
- TNF Alpha Blocker: Patients with skin diseases taking TNF alpha blockers
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteer | Azathioprine | TNF Alpha Blocker | Total
Number analyzed (Participants) | 21 | 10 | 12 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 9 | 12 | 42
  >=65 years | 0 | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (9.5) | 57 (7.3) | 40 (11.6) | 38.1 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 7 | 3 | 23
  Male | 8 | 3 | 9 | 20
Region of Enrollment [Number; unit: participants]
  United States | 21 | 10 | 12 | 43

OUTCOME MEASURES:

1. Primary Outcome: Influenza Hemagluttination Inhibition Titers Measured Against H3N2 Perth Before and After Influenza Vaccination
Description: Influenza hemagluttination inhibition titers were measured against H3N2 Perth before and after influenza vaccination. Titers greater than or equal to 1:40 constitute a protective response to influenza strains.
Time Frame: 28 days
Measure: Number; unit: participants
Groups:
- TNF Alpha Blockers: Patients with skin diseases taking TNF alpha blockers
Arm/Group | Healthy Volunteer | Azathioprine | TNF Alpha Blockers
Number analyzed (Participants) | 21 | 10 | 12
participants | 19 | 5 | 6

2. Primary Outcome: Influenza Hemagluttination Inhibition Titers Measured Against Pandemic H1N1 Strains Before and After Influenza Vaccination
Description: Influenza hemagluttination inhibition titers were measured against pandemic H1N1 strains before and after influenza vaccination. Titers greater than or equal to 1:40 constitute a protective response to influenza strains.
Time Frame: 28 days
Measure: Number; unit: participants
Arm/Group | Healthy Volunteer | Azathioprine | TNF Alpha Blockers
Number analyzed (Participants) | 21 | 10 | 12
participants | 15 | 3 | 6

ADVERSE EVENTS:
Groups:
- Healthy Volunteer Pre-vaccination: Healthy volunteers who had blood drawn prior to vaccination with influenza vaccine
- Healthy Volunteer Post-vaccination: Healthy volunteers who had blood drawn after vaccination with influenza vaccine
- Azathioprine Pre-vaccination: Patients with skin disease treated with azathioprine who had blood drawn prior to vaccination with influenza vaccine
- Azathioprine Post-vaccination: Patients with skin disease treated with azathioprine who had blood drawn after vaccination with influenza vaccine
- TNF Alpha Blocker Pre-vaccination: Patients with skin disease treated with TNF blockers who had blood drawn prior to vaccination with influenza vaccine
- TNF Alpha Blocker Post-vaccination: Patients with skin disease treated with TNF blockers who had blood drawn after vaccination with influenza vaccine
Arm/Group | Healthy Volunteer Pre-vaccination | Healthy Volunteer Post-vaccination | Azathioprine Pre-vaccination | Azathioprine Post-vaccination | TNF Alpha Blocker Pre-vaccination | TNF Alpha Blocker Post-vaccination
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/10 | 0/10 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/10 | 0/10 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No